CLINICAL TRIAL: NCT03227510
Title: Circulating MicroRNAs as Biomarkers in Hepatocellular Carcinoma Among Somali Patients
Brief Title: MicroRNAs as Diagnostic Biomarkers in Hepatocellular Carcinoma Among Somali Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: People's Friendship University of Russia (Other)
Responsible Party: Principal Investigator, Mohamed Abdulkadir Hassan, MD, People's Friendship University of Russia
Other Study IDs: 1072178049
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma , MicroRNAs, Somalia
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sample from patients with HCC and from chronic liver disease and healthy volunteer controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HCC Cases (Group 1): This group will include 63 subjects and the diagnoses will be based on clinical examination, laboratory tests such as (Liver Function tests, Alpha-fetoprotein , Ultrasound, and biopsy in some cases if possible (Depends on the patients and their financial issues).
- Chronic Liver Diseases (group 2): This group will be including 31 patients, and the diagnoses will be based on laboratory such as (liver function tests, viral markers, AFP,) and by ultrasound findings (shrunken liver, coarse echo-pattern, attenuated hepatic vein and finding nodular surface)
- Healthy Volunteer (group 3): It will include 32 subjects that serve as control group.
  These all patients and control groups will be subject the following parameters: Biochemical tests such as (Liver function tests, viral markers, serum AFP, CBC, Kidney functions and others) and circulating MicroRNAs levels of all these subjects.

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer and is the third leading cause of cancer that related death in the worldwide. Although, current most of doctors and laboratorians of HCC diagnoses bases are medical imaging such ultrasound, MRI, CT-scan and laboratory analyses tests for serum tumor markers such as alpha-fetoprotein (AFP) which characterized by very low of sensitivity in the detection of HCC. Last two decades, scientists was focused researches of small molecules called MicroRNAs which are produced by human cells and can be released in the blood.

MicroRNAs are class of (20 - 25 nucleotide in length) non-coding RNAs, and its emerging non-invasive diagnostic biomarker for cancer diagnosing, screening, monitoring treatment and to predict prognosis. A number of studies exposed an abnormal expression of human serum MicroRNAs in many tumors such as liver, pancreatic and colorectal carcinoma. Recently, MicroRNAs have a role in the development of HCC, but still it is unknown if these small molecules will be used as biomarker for diagnosis and survival of HCC.

The aim of this study is to establish MicroRNAs as biomarkers for diagnostic tool of HCC patients and to compare to circulating levels of MicroRNAs in chronic liver diseases patients and health volunteers and those HCC patients and To determine the clinical utility of MicroRNAs as a diagnostic maker of hepatocellular carcinoma comparing with alpha fetoprotein the current marker of (HCC).

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer and is the third leading cause of cancer that related death in the worldwide. According the burden of cancer in economically developing countries is increasing in a result of population aging and growth in addition to increasing the adaptation of cancer-related lifestyle choices such as physical inactivates, smoking and western diets. Liver cancer in women are seventh most common diagnosed cancer and sixth most cause of cancer death while in men are fifth diagnosed cancer and second cause of cancer death. In 2008 liver cancer new cases were estimated 748,300 and death cases were 695,900 occurred in worldwide. Viral hepatitis infections, alcohol, fungal toxins (aflatoxins), food additives, toxins produced industrial chemicals and water and air pollutants are the major factors of primary liver cancer.

Although, current most of doctors and laboratorians of HCC diagnoses bases are medical imaging such ultrasound, MRI, CT-scan and laboratory analyses tests for serum tumor markers such as alpha-fetoprotein (AFP) which characterized by very low of sensitivity in the detection of HCC. Last two decades, scientists was focused researches of small molecules called MicroRNAs which are produced by human cells and can be released in the blood.

MicroRNAs are class of (20 - 25 nucleotide in length) non-coding RNAs, and its emerging non-invasive diagnostic biomarker for cancer diagnosing, screening, monitoring treatment and to predict prognosis. A number of studies exposed an abnormal expression of human serum MicroRNAs in many tumors such as liver, pancreatic and colorectal carcinoma. Recently, MicroRNAs have a role in the development of HCC, but still it is unknown if these small molecules will be used as biomarker for diagnosis and survival of HCC.

Purpose:

1. To recognize serum microRNAs as a diagnosis or prediction biomarker for Hepatocellular carcinoma.
2. To correlate with the expression level of microRNAs between HCC patients , chronic liver disease and health volunteer subjects.
3. To determine the clinical utility of MicroRNAs as a diagnostic maker of Hepatocellular carcinoma comparing with alpha fetoprotein the current marker of (HCC).

Methods Study design: This is observational study (Case Control Study). A total of 126 subjects aged over 18 years old; that divided into three groups will be enrolled in this study in Dufle Specialist Hospital; these groups are HCC group, Chronic liver disease group and health volunteer group. The diagnosed criteria of HCC group are ultrasound which its nodules more than 5cm, liver function tests, viral markers and AFP. The other groups (chronic liver disease and health) the diagnoses will be based on laboratory such as (liver function tests, viral markers, AFP, complete blood count (CBC), Kidney functions and others) the clinical and laboratory analysis data will be collected perceptively The blood samples will be collected at one time, after that the blood samples will be separated using Serum-separating tubes and then centrifuges to get the serum and will be stored in -20°C before transferred from Somalia to Russia.

Viral marker Hepatitis B surface antigen (HBsAg) and antibody to HCV (anti-HCV) will be checked using commercially available enzyme linked immunosorbent assay kits for every subject of these three groups.

The expression of MicroRNAs will be detected by quantitative reverse-transcriptase polymerase chain reaction (qRT-PCR) with human TaqMan MicroRNA Assay Kits (Applied Biosystems) of these groups either HCC group , Chronic liver disease and healthy volunteers. The investigators will define the groups of HCC, Chronic liver disease and healthy volunteers with high or low expression based on the median expression value of each microRNA.

All statistical analyses will be carried out with Statistical Package for the Social Sciences (SPSS) version 20. MicroRNAs expressions among different group (HCC, Chronic liver diseases, and healthy volunteers) will be analyzed by SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HCC patients through history taking and physical Examination, AFP and ultrasonography (> 5cm in size).
* Chronic liver disease patients with history of liver disease rather than HCC such as cirrhosis, chronic viral hepatitis, non-alcoholic liver disease (NALD).
* Healthy volunteers with no history of liver problems.
* Informed consent from all participants before enrollment in the study.

Exclusion Criteria:

* HCC less than 5 cm in size during ultrasound examinations
* Extrahepatic disease, other primary tumour
* Inability to provide informed consent or who refused to draw off blood.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be carried out on 126 subjects who will be admitting from the outpatient clinic of Dufle Specialist Hospital Mogadishu, Somalia.
  They will be classified into 3 groups:
  Group I: It will include 63 HCC subjects. Group II: It will include 31 chronic liver disease patients. Group III: It will include 32 healthy volunteer subjects
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
MicroRNAs and its Correlation to Development and prediction of HCC | 6 months to 1 year
  Circulating MicroRNAs levels in serum samples from HCC, Chronic liver diseases and health volunteers Somali subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel P Ogurtsov, MD, Study Chair — People's Friendship University of Russia; Mohamed A Hassan, Principal Investigator — RUDN University, Abrar University

IPD SHARING:
Plan to Share IPD: No